CLINICAL TRIAL: NCT04656405
Title: Evaluation of Efficacy of Online Real-time Quality Measurement and Feedback Video-based CPR Training Program
Brief Title: Efficacy of Online Real-time CPR Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Han Kim, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 30-2020-232
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Cardiopulmonary Resuscitation; Education
Keywords: Cardiopulmonary Resuscitation; Education; Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online real-time CPR training program (Experimental): Online real-time quality measurement and feedback video-based CPR training will be provided to participants
  Interventions: Other: Online real-time quality measurement and feedback video-based CPR training
- Online real-time CPR training without quality measurement program (Active Comparator): Online real-time feedback video-based CPR training without quality measurement will be provided to participants
  Interventions: Other: Online real-time feedback video-based CPR training without quality measurement
- Conventional CPR training program (Placebo Comparator): Conventional CPR training will be provided to participants
  Interventions: Other: Conventional CPR training

INTERVENTIONS:
Other: Online real-time quality measurement and feedback video-based CPR training — Participants in the online real-time quality measurement and feedback video-based CPR training program group will access an online training center with laptop computers provided by the researcher. All education and communication is conducted online. The study instructors shows the study participants an edited version of the CPR training video used in the conventional CPR training program. A Little Anne QCPR mannequin (Laerdal, Stavanger, Norway) and SkillGuide (Laerdal, Stavanger, Norway) are provided so that the participants can use while watching the video and during the following hands-on practice session.
  After watching the video, hands-on practice will be conducted by the instructor on-line. The instructor will watch each individual participants CPR performance via video conferencing and collect real-time performance data using the QCPR mannequin device. Using this information, the instructor will provide real-time online feedback to participants.
  Arms: Online real-time CPR training program
Other: Online real-time feedback video-based CPR training without quality measurement — Participants in the online real-time feedback video-based CPR training without quality measurement program group will access an online training center with laptop computers provided by the researcher. All education and communication is conducted online. When study participants access the online training center, study instructors shows the study participants an edited version of the CPR training video used in the conventional CPR training program. A Little Anne QCPR mannequin (Laerdal, Stavanger, Norway) is provided so that the participants can use while watching the video and during the following hands-on practice session.
  After watching the video, hands-on practice will be conducted by the instructor on-line. The instructor will watch each individual participants CPR performance via video conferencing. The instructor will provide real-time online feedback to participants.
  Arms: Online real-time CPR training without quality measurement program
Other: Conventional CPR training — Participants in the conventional CPR training program group will be provided CPR education with the "Home Education and Resuscitation Outcome Study (HEROS)" program that is currently provided in Seoul, Korea. The HEROS program is a 1-hour training course, consisting of a 30-minute video-based self-instruction training with a mannequin. The program also includes a bystander CPR simulation with a simulated dispatcher using the participants own cell phone. Little Anne QCPR mannequin (Laerdal, Stavanger, Norway) and SkillGuide (Laerdal, Stavanger, Norway) device are provided to measure and give feedback on the participants CPR performance.
  Arms: Conventional CPR training program

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a new online real-time quality measurement and feedback video-based CPR training program. The study participants will be allocated to three different CPR training programs: online real-time quality measurement and feedback video-based CPR training program, online real-time feedback video-based CPR training without quality measurement program, and conventional CPR training program. After CPR training, each participant will perform a 6 minute CPR simulation test. The investigators will compare the quality of chest compression between the three study groups. The investigators hypothesize that the new online real-time quality measurement and feedback video-based CPR training program is non-inferior to the preexisting conventional CPR training program and is superior to online real-time feedback video-based CPR training without quality measurement.

DETAILED DESCRIPTION:
Bystander CPR is important for the survival of out-of-hospital cardiac arrest patients. CPR training for the general public is important to improve the rate and quality of bystander CPR. Preexisting CPR education was conducted under face-to-face contact with instructors and multiple trainees gathering at a training center, but after the coronavirus disease 2019 pandemic, face-to-face training became difficult. To overcome this limitation the investigators have developed a new online real-time quality measurement and feedback video-based CPR training program that uses online video conferencing, Little Anne QCPR mannequin (Laerdal, Stavanger, Norway) and SkillGuide (Laerdal, Stavanger, Norway) device.

The purpose of this study is to evaluate the effectiveness of a new online real-time quality measurement and feedback video-based CPR training program. To evaluate the effectiveness of the new CPR training program the investigators propose to conduct a randomized clinical trial with three arms: online real-time quality measurement and feedback video-based CPR training program, online real-time feedback video-based CPR training without quality measurement program, and conventional CPR training program. 60 non healthcare provider, healthy adult volunteers will be randomized to each study arm. After CPR training, each participant will perform a 6 minute CPR simulation test. The investigators will measure the depth and rate of chest compression, hand positioning during chest compression, no-flow time and start to chest compression time.

The primary outcome of the study is mean chest compression depth. Chest compression rate, hand position, total no flow time, and time to chest compression will also be measured. The investigators hypothesize that the new online real-time quality measurement and feedback video-based CPR training program is non-inferior to the preexisting conventional CPR training program and is superior to online real-time feedback video-based CPR training without quality measurement.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 18 years or older

Exclusion Criteria:

* Healthcare providers
* Participants with chronic lung diseases
* Participants with cardiovascular diseases
* Participants with visual disabilities
* Participants with hearing disabilities
* Participants with musculoskeletal disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Chest compression depth | Assessed during 6 minute CPR simulation test
  Depth of chest compressions measured in millimeters

SECONDARY OUTCOMES:
Chest compression rate | Assessed during 6 minute CPR simulation test
  Rate of chest compression per minute
Hand position | Assessed during 6 minute CPR simulation test
  Correct hand position measured by QCPR mannequin
No flow time | Assessed during 6 minute CPR simulation test
  Time with no chest compression after start of chest compression
Time to chest compression | Assessed during 6 minute CPR simulation test
  Time from start of simulation to start of chest compression

CONTACTS AND LOCATIONS:
Overall Officials: TAE HAN KIM, MD, Study Chair — SMG-SNU Boramae Medical Center; STEPHEN GW LEE, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul Metropolitan Government-Seoul National University Borame Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim TH, Lee YJ, Lee EJ, Ro YS, Lee K, Lee H, Jang DB, Song KJ, Shin SD, Myklebust H, Birkenes TS. Comparison of Cardiopulmonary Resuscitation Quality Between Standard Versus Telephone-Basic Life Support Training Program in Middle-Aged and Elderly Housewives: A Randomized Simulation Study. Simul Healthc. 2018 Feb;13(1):27-32. doi: 10.1097/SIH.0000000000000286. PMID 29369963
- [Background] Park GJ, Kong SYJ, Song KJ, Shin SD, Kim TH, Ro YS, Myklebust H, Birkenes TS. The Effectiveness of a New Dispatcher-Assisted Basic Life Support Training Program on Quality in Cardiopulmonary Resuscitation Performance During Training and Willingness to Perform Bystander Cardiopulmonary Resuscitation: A Cluster Randomized Controlled Study. Simul Healthc. 2020 Oct;15(5):318-325. doi: 10.1097/SIH.0000000000000435. PMID 32604135
- [Background] Cheng A, Nadkarni VM, Mancini MB, Hunt EA, Sinz EH, Merchant RM, Donoghue A, Duff JP, Eppich W, Auerbach M, Bigham BL, Blewer AL, Chan PS, Bhanji F; American Heart Association Education Science Investigators; and on behalf of the American Heart Association Education Science and Programs Committee, Council on Cardiopulmonary, Critical Care, Perioperative and Resuscitation; Council on Cardiovascular and Stroke Nursing; and Council on Quality of Care and Outcomes Research. Resuscitation Education Science: Educational Strategies to Improve Outcomes From Cardiac Arrest: A Scientific Statement From the American Heart Association. Circulation. 2018 Aug 7;138(6):e82-e122. doi: 10.1161/CIR.0000000000000583. PMID 29930020
- [Background] Baldi E, Cornara S, Contri E, Epis F, Fina D, Zelaschi B, Dossena C, Fichtner F, Tonani M, Di Maggio M, Zambaiti E, Somaschini A. Real-time visual feedback during training improves laypersons' CPR quality: a randomized controlled manikin study. CJEM. 2017 Nov;19(6):480-487. doi: 10.1017/cem.2016.410. Epub 2017 Jan 24. PMID 28115027